CLINICAL TRIAL: NCT05341973
Title: The Effect of Self-efficiency Support Given to Hypertension Patients on the Patients' Disease Management and Self-management Levels
Brief Title: The Patients' Disease Management and Self-management Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bahar Ciftci, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/55
Record Dates: First submitted 2022-04-13; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): The Self- Management Program Developed will increase Self-Efficacy, Self-Care Management in Hypertension Patients.
  Interventions: Behavioral: Education
- Control (No Intervention): It will not change the Self-Efficacy, Self-Care Management in Hypertension Patients of the Self-Management Program.

INTERVENTIONS:
Behavioral: Education — Self-Management Program will increase Self-Efficacy, Self-Care Management in Hypertension Patients.
  Arms: Education

SUMMARY:
The purpose of this research; The aim of this study is to examine the effects of self-management support given for hypertension patients on patients' adherence to treatment and disease, self-efficacy level, self-care management. This research is a randomized controlled and pretest-posttest applied design. The research will be carried out in Van Yüzüncü Yıl University Research Hospital with patients previously diagnosed with hypertension. The population of the research will consist of patients who have previously applied to the hospital where the research will be conducted and who have been diagnosed with hypertension who meet the research criteria. After the power analysis, it is planned to include 150 hypertension patients in the sample of the study. All patients in the intervention and control groups who meet the inclusion criteria will be verbally informed about the purpose of the study and the method of application, and their consent will be obtained. The pretest forms required for the research will be filled in by face-to-face interview method for all patients. In the study, the number of individuals in the randomization group will be determined by using the computer program, provided that they are equal in number. All materials prepared for self-management support will be delivered to the patients in the intervention group and they will be taught how to use them by the demonstration method. Patients will be asked to do the same procedure and the process will continue until they ensure correct use. Participants will be informed that there is a phone number that they can call whenever they want, when there are subjects that are not understood or that need to be repeated. Patients will be called three times a week and necessary checks will be made on blood pressure monitoring, nutrition, weight control, etc. In this way, patients in the intervention group will be followed remotely by tele-nursing for 3 months, their questions will be answered when they encounter problems, and guidance will be given in case of emergency. No intervention will be made in the control group. Necessary forms will be re-administered to all patients in both groups after 3 months as a post-test. At the end of the research, a comparison of the intervention and control groups will be made.

DETAILED DESCRIPTION:
Type of research This project is a randomized controlled and pretest- posttest applied design. Location and Characteristics of the Research The research will be carried out in Van SBU Training and Research Hospital Research Hospital with patients who have been diagnosed with hypertension before.

The number of cardiology outpatient clinics of Van Training and Research Hospital is 5. In our hospital, there are cardiology and internal departments that also include hypertension patients. There are 70 patients per day per cardiology outpatient clinic. The majority of them are individuals with hypertension and hypertension, as well as additional chronic diseases. It is questioned whether individuals follow their weight, whether they change their eating and drinking habits, whether they use their medications regularly, and finally whether they follow their blood pressure regularly. After this questioning, examination and various tests (blood analysis, ultrasound, etc.), the medicines of the patients are regulated. In general, patients are called for control every 2 months. However, this period is extended for individuals who take the warnings into account, measure their blood pressure regularly and see that it is stable at the expected level.

Research Population and Sample Selection The population of the research will consist of patients who have previously applied to the hospital where the research will be conducted and who have been diagnosed with hypertension who meet the research criteria.

The sample was calculated using the Hill-Bone Hypertension Treatment Adherence Scale, which was used in 2 studies (51.52). In order to determine the sample size, a priori power analysis was performed and it was determined that at least 55 hypertension patients were required for each of the intervention and control groups in order for the power of the study to exceed 80% at the 95% confidence interval, 0.05 significance level and medium effect size ( 50). In case of data loss, a total of 150 data will be collected by including 10% backup sample to this number. After the posttest data are collected, the power analysis will be looked at again. In the final power analysis, this rate is expected to exceed 90%.

For sampling calculation, Hill-Bone Hypertension Treatment Adherence Scale was used (51-52).

Inclusion criteria for the study:

Follow-up for at least 6 months with the diagnosis of essential hypertension, Using antihypertensive drugs, No change in antihypertensive drug treatment in the last 1 month, Not having any other accompanying chronic disease (Diabetes mellitus, cancer, chronic kidney failure, chronic obstructive pulmonary disease, heart failure, etc.), Having no mental or communication problems, Computer/tablet/smartphone etc. to watch videos. having technological tools, Having internet, Being over 18 years old, Having at least primary education level, Not being pregnant or lactating, Data collection tools and features The data of the research; Patient Information Form, Hill-Bone Hypertension Treatment Adherence Scale, Self-Care Management Scale in Chronic Diseases, 6-item Self-Efficacy for Managing Chronic Diseases (SEMCD6) Scale, Chronic Disease Adherence Scale (CHUS), and Patient Education Satisfaction Scale (HEMÖ), Hypertension Management Information Booklet will be collected using Hypertension Management Video CDs.

Data Collection All patients in the intervention and control groups who meet the inclusion criteria will be verbally informed about the purpose of the study and the method of application. "Informed Consent Form" will be filled in for the patients who agree to participate in the study. Then, the pre-test forms will be filled in by face-to-face interview method for all patients in the intervention and control groups.

In the study, "stratification and block randomization methods" will be used in assigning participants to control and intervention groups. In the literature, it has been reported that age, gender and educational status are among the factors affecting drug and disease compliance, self-efficacy and self-management of hypertension patients. In line with this information, "age, gender and educational status" variables will be used in the stratification of hypertension patients in the study. Accordingly, patients will be stratified as "18-40, 41-60, 61 and above" for the age variable, "female and male" for the gender variable, "Primary School, Secondary School, High School and above" for the educational status variable, and randomization with blocks will be applied. In addition, 75 hypertension patients will be included in each of the study groups by ensuring that the layers are repeated five times in the study (2X2X2X5).

Enterprise Group; All materials prepared for Self-Management Support will be delivered to the patients and they will be taught how to use them by the demonstration method. Patients will be asked to do the same procedure and will continue to be taught until they use it correctly. Participants will be informed that there is a phone number that they can call whenever they want, when there are subjects that are not understood or that need to be repeated.

Phone; All patients will be registered on the telephone line to be used by the researchers and the telephone will be used only for research. The phone will be available at the cardiology nurse Sümeyra Autonomous. When the cardiology nurse Sümeyra Özerk could not be reached, so that the patients are not victims and that they can reach the phone whenever they want, the project coordinator Dr. Instructor A phone call will be made to member Bahar Çiftçi. At the same time, a group with the entire project team will be established and the arrangements for the project will be discussed there.

Management of hypertension, ability to measure blood pressure at home, edema control, nutrition, movement, salt restriction, etc. Self- management support will be provided by providing training to teach. Patients will be called three times a week and necessary controls will be provided on training, blood pressure monitoring, nutrition, weight control, etc. It will be required to measure and record blood pressure twice a day with a digital and easy-to-use sphygmomanometer. In addition, it will be reminded that height-weight, blood pressure should be measured and recorded. It will be ensured that the materials sent to the patients are used in the measurement of height, weight and blood pressure. Patients will be reminded that they need to take measurements twice a day, and they will be warned to call the phone number that they can reach in case of emergency if an abnormal situation is encountered. In this way, patients in the intervention group will be followed remotely by tele-nursing for 3 months, their questions will be answered when they encounter problems, and guidance will be given in case of emergency.

The content of the videos will be the same as the Training Booklet. The videos are planned to be between 3-5 minutes. It is planned to have videos that are explained in simple language that patients can understand. In addition, the videos will be presented to the patient after review. In the inclusion criteria of the research, "Computer/tablet/smartphone etc. to watch the videos. The videos can be watched comfortably, as it is a requirement to have "technological tools". Patients in the intervention group will be able to access the videos whenever they want. The videos will be shared only with the patients in the intervention group throughout the research. When the data collection phase is over, the videos will be shared first with the control group and then on the social media platform that hypertension patients can access.

Evaluation of data The data will be evaluated in the SPSS (Statistical Package for Social Sciences for Windows, Version 22.0) package program. In the evaluation of the data, the statistical significance value will be accepted as 0.05, the Type 1 error will be kept at 5% and the evaluation will be made with a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up for at least 6 months with the diagnosis of essential hypertension,
* Using antihypertensive drugs,
* No change in antihypertensive drug treatment in the last 1 month,
* Not having any other accompanying chronic disease (Diabetes mellitus, cancer, chronic -kidney failure, chronic obstructive pulmonary disease, heart failure, etc.),
* Having no mental or communication problems,
* Computer/tablet/smartphone etc. to watch videos. having technological tools,
* Having internet,
* Being over 18 years old,
* Having at least primary education level, Not being pregnant or lactating,

Exclusion Criteria:

* Follow-up for less than 6 months with the diagnosis of essential hypertension,
* Not using antihypertensive drugs,
* Changes in antihypertensive drug therapy in the last 1 month,
* Presence of another concomitant chronic disease (Diabetes mellitus, cancer, chronic -kidney failure, chronic obstructive pulmonary disease, heart failure, etc.),
* Having a mental or communication problem,
* Computer/tablet/smartphone etc. to watch videos. lack of technological tools,
* Lack of internet,

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Self-Care Management Scale in Chronic Diseases (KHÖBYÖ) | 3months
  he scale consists of 35 items and is in a five-point Likert type (1 = strongly disagree, 2 = disagree, 3 = undecided, 4 = agree, 5 = strongly agree). Self- protection (items 2, 6, 8, 11, 15, 18, 19, 20, 22, 23, 25-34), and social protection (1, 3, 4, 5, 7, 9, 10, 12) There are two sub-dimensions (items 13, 14, 16, 17, 21, 24 and 35). Items 3, 15, 19 and 28 in the scale are negative statements. The total scores that can be obtained from the scale vary between 35-175 points, and an increase in the score indicates that the individual's self-care management also increases.
The 6-item Self-Efficacy for Managing Chronic Diseases Scale(SEMCD6) | 3months
  It is an easy-to-use and effective tool for assessing the self-efficacy levels of patients with chronic diseases. The scale is rated on a 10-point scale ranging from "not at all sure" to "very sure". The score obtained from the scale is the average of 6 items, and high scores indicate high self-efficacy. If more than 1 answer is given to an item and the items are consecutive, the low score is included in the calculation. If the 2 answers given are not consecutive, this item is excluded from the calculation. In order for the scale to be calculated, at least 4 items must be answered.

CONTACTS AND LOCATIONS:
Overall Officials: BAHAR Çiftçi, Study Director — Ataturk University
Locations (1):
- BAHAR Çiftçi, Erzurum, Turkey (Türkiye)